CLINICAL TRIAL: NCT07065708
Title: Transperineal Ultrasound as a Biofeedback Tool for Pelvic Floor Muscle Therapy in Postpartum Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Rahim Asad Abdul, Staff Physician, Singapore General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-4537
Record Dates: First submitted 2025-06-25; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Pelvic Floor Muscle Training; Transperineal Ultrasound; Biofeedback Therapy; Postpartum; Pelvic Floor Disorder; Pelvic Floor Muscle Exercise; Pelvic Floor, Obstetric; Pelvic Floor Dysfunction; Pelvic Floor Health After Childbirth; Physiotherapy; Physiotherapy Specialty
Keywords: pelvic floor muscle training; biofeedback; transperineal ultrasound; pelvic floor exercises; physiotherapy; pelvic floor dysfunction; pelvic floor disorder; pelvic floor contraction
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): Participants will receive tranperineal ultrasound scan but will not receive visual biofeedback (i.e. they will not be able to see images of their pelvic floor when attempting to perform pelvic floor muscle contractions)
  Interventions: Diagnostic Test: Transperineal ultrasound without visual biofeedback
- Study Arm (Experimental): Participants will receive tranperineal ultrasound scan with visual biofeedback
  Interventions: Diagnostic Test: Visual biofeedback using transperineal ultrasound

INTERVENTIONS:
Diagnostic Test: Visual biofeedback using transperineal ultrasound — Transperineal ultrasound with visual biofeedback
  Arms: Study Arm
Diagnostic Test: Transperineal ultrasound without visual biofeedback — Transperineal ultrasound without visual biofeedback
  Arms: Control Arm

SUMMARY:
Regular and effective pelvic floor muscle exercises after vaginal birth are crucial in reducing the risk of pelvic floor disorders in women. Pelvic floor muscle exercises are generally encouraged by healthcare providers to their patients after birth. However, it is often difficult to confirm whether a patient is performing pelvic floor muscle contractions correctly. A supervised pelvic floor physiotherapy session allows a professional to assess the pelvic floor and give their verbal feedback to patients. However even in this setting, patient's are reliant on the physiotherapist and have no way to assess their own performance. The 'biofeedback approach' allows for the clinician and patient to visually assess and modify their performance and can potentially allow for more effective therapy and better engagement. Transperineal ultrasonography is a widely available, safe and non-invasive biofeedback tool that can used at the bedside in order to assess pelvic floor muscle contractions. Our aim is to assess if using transperineal ultrasound can enhance the ability of postpartum patients to perform effective pelvic floor muscle therapy.

DETAILED DESCRIPTION:
This is a prospective, randomised controlled study and will be conducted through five stages:

Stage 1: Recruitment and randomisation. Stage 2: Assessment. Stage 3: Preliminary analysis and Interim report. Stage 4: Follow up assessment. Stage 5: Final analysis.

Stage 1: Recruitment and Randomisation Postpartum patients who attend the pelvic floor assessment clinic will be screened for eligibility to the study. The study team will be responsible for screening and recruiting the participants based on the aforementioned inclusion/exclusion criteria. If eligible, the potential participant will be approached by a member of the study team and provided with a Participant Information Sheet and Consent Form. If they agree, they will be recruited to the study and will be allocated a study identifier number (SIN). A memberof the study team will take written consent from the participant. English will be the default language of use; however, interpretation will be available in both Chinese, Malay and Tamil if required. Participants will be randomized into two different arms for the study (control arm and study arm). Each participant will be asked to complete the pre-study questionnaire. Equal numbers are required in each arm and therefore randomization will be performed using a computer randomizer set to distribute SINs into two equal groups.

Stage 2: Assessment Assessment of participants is divided into two parts. The first part involves the gathering of clinical data such as demographic, pregnancy, and symptom information. This is obtained through their electronic medical record (using only the Citrix application), as well as eliciting symptoms history verbally from the participant. A clinical examination for uterovaginal prolapse is performed and a digital examination to assess pelvic floor muscle tone, known as the Modified Oxford Scale (MOS), is recorded in the standing position. This assessment forms part of the usual care for each of the participants and can therefore be performed by any qualified member of their clinical care team. After this assessment, study participants are provided with a specially designed hard-copy questionnaire to complete which is relevant to the aims of the study. This is to ascertain the participants knowledge of, and exposure to pelvic floor muscle therapy. The second part of the assessment is conducted by a member of the study team specialized in transperineal ultrasound of the pelvic floor and pelvic floor muscle training techniques. Each participant is asked to undress from the waist down and lay supine for the examination. A chaperone is present and dignity is maintained throughout. Participants will be encouraged to "squeeze the muscles" of their perineum and several attempts will be given to each participant to achieve this. Verbal feedback will be given by the assessor after each attempt to be sure the participant is activating their pelvic floor muscles and not co-activating their abdominal or gluteal muscles. Transperineal ultrasound is then performed for all participants. Preparation of the probe involves applying a single-use, non-latex probe cover around a GE™ RAB2-5-MHz 3-dimensional volume transducer with generous amounts of ultrasound conducting gel placed inside and outside the probe cover. The transducer is placed upon the participant's perineum, in the mid-sagittal plane, and acquisition of images in conducted through a Voluson™ S10 ultrasound system. An acquisition angle of 85° is set and the machine is configured to the "Pelvic Floor" setting. Participants in the control arm will have the ultrasound screen turned away from them with only the assessor having access to it. One 3dstatic image of the pelvic floor at rest will be obtained. The assessor will then ask the participant to perform a pelvic floor muscle contraction where a 4d dynamic image of the pelvic floor will be obtained. Three attempts at pelvic floor muscle contraction will be made for each participant. During this time the assessor will provide no feedback nor encouragement to the participant. Participants in the study arm will have the ultrasound screen turned towards them in a way that both the assessor and participant can view it. A simple demonstration of the pelvic anatomy will be given to the participant outlining the orientation of the image as well as the basic pelvic structures such as positions of the bladder, vagina and rectum. As in the control group, the assessor will obtain the same static 3d image of the pelvic floor at rest as well as three dynamic 4d images during a pelvic floor contraction. Unlike the control group, the participant will be able to visualize in real-time the dynamic movement of their pelvic floor. They will be permitted to adjust/strengthen their technique between attempts based on these visual cues. Upon completion of the assessment, all participants will have a follow up visit arranged in 3 months. This appointment usually forms a standard part of their clinical care and will be utilized to perform the follow up assessment. Participants who wish to continue to take part in the study will be informed that they will have the opportunity to repeat the assessment again during their follow up visit and will be encouraged to continue to perform pelvic floor muscle therapy in the interim.

Stage 3: Preliminary analysis and Interim report This stage is performed by the study team only and does not require the involvement of the participants. Ultrasound data sets will be evaluated by a member of the study team who is blinded to the clinical data as well as to the study arm that the data set belongs to. The following describes the measurement parameters which are relevant to the study. a. Antero-posterior (AP) pelvic hiatal diameter. This is defined as the distance between the inferior edge of the symphysis pubis and the greatest apogee of the puborectalis muscle. The measurement can be obtained in both the mid-sagittal as well as the transverse (axial) plane. However, care must be taken to orientate the 3d/4d image to reflect the correct plane of viewing regardless of the method of measurement. It is well established that the AP hiatal diameter is a very good indicator of pelvic floor muscle contraction. Based on a previous study, a proportional change in AP hiatal diameter of >15% corresponds well with a normal pelvic floor muscle contraction. This cut-off value will be utilized to determine the adequacy of contraction. b. Transverse diameter This is defined as the maximal diameter between the inner edge of the levator ani muscles and is measured solely in the transverse plane. As with AP diameter, changes in transverse diameter are associated with effective muscle contractions, albeit to a lesser extent. The transverse diameter can be a useful adjunct to the AP diameter as it provides assurance that that a pelvic floor contraction is effective. c. Pelvic hiatal area This is the defined as the area enclosed anteriorly by the symphysis pubis, laterally by the levator ani and posteriorly by the puborectalis. This measurement can only be obtained in the transverse plane and conventionally measured along the axis subtended by the symphysis pubis and greatest apogee of the puborectalis. Changes in the pelvic hiatal area correspond well with clinical assessments, such as use of the MOS. Care will be taken to ensure the correct plane is measured during rest and contraction and measurement of the area will be performed by tracing the inner outline using the trace function on the Voluson™ S10 ultrasound system. Preliminary analysis will be performed when the minimal sample size has been reached. Results of the analysis will form the basis of the studies' interim report. The interim report will ultimately aim to answer the primary hypothesis of the study- to determine if a significant difference is observed in pelvic floor muscle contraction between the study group and the control group. However, prior to this, several quality assurance checks will be performed. These quality assurance measures are described later. The interim report will also explore if there were any issues/adverse effects of the study and if so, whether this would warrant discontinuation of the trial. The investigators do not anticipate any adverse physical effects of the study as the use of ultrasound is very safe. However, the investigators do anticipate that some participants within the control group may wish to visualize their pelvic floor anatomy on ultrasound. As this would compromise the validity of the next stage of the study, the investigators would be required to withdraw the participant from the study at this stage if they were to request this. The investigators would be able to grant this request willingly at the end of the next stage as visualization after Stage 4 is complete will not compromise the results of the study.

Stage 4: Follow up assessment This stage will occur 3 months after the initial assessment stage. Participants enrolled in the study will be invited back for a follow up review consisting of an assessment of any symptoms, adherence to PFMT and repeat ultrasound assessment of their pelvic floor muscle strength. As previously mentioned, the follow up stage is part of the standard clinical care for each patient and therefore the study will be done in parallel with their usual clinical care. Asimilar method of assessment will be employed to the initial assessment, where a physical examination for uterovaginal prolapse and MOS grading are conducted. TPUS assessment will be done at rest, but when performing a pelvic floor muscle contraction, all participants will be blinded from visual biofeedback. Only the assessor will have access to the ultrasound screen and no verbal feedback or encouragement will be given during this time. As with the initial assessment three attempts at pelvic floor muscle contraction will be given to each participant with the best one being used for final analysis. The assessors themselves will be blinded to clinical data as well as the results of the previous assessment. Data will continue to be de-identified, using only the SIN as a reference to data sets. The follow up will also be an opportunity to address any adverse effects or difficulties each participant may have experienced since the initial assessment. These will be thoroughly documented as part of the study results and will be managed appropriately by their clinical care team. The CIRB will be informed of any adverse event the participant suffers as a result of their participation in the study. Participant involvement will end at this stage. If requested, participants in the control arm, may view the images of the pelvic floor at rest and during contraction. Advice will be given to them on how to manage their pelvic floor symptoms and an opportunity for questions will be provided. Each participant will be encouraged to complete a post-study questionnaire outlining their experiences.

Stage 5: Final analysis The objective of the final analysis will be to assess if both the primary and secondary outcomes have been met. As with the preliminary analysis, participants are not required at this stage. Measurements of validated parameters will be obtained from each data set (initial and 3-month follow up) from each participant. These measurements as well as will be compared between time periods to assess if (a) postpartum patients continue to perform PFE; (b) are they still effective; and (c) is visual biofeedback more useful than no biofeedback.

ELIGIBILITY:
Inclusion Criteria:

* Female participants
* Aged 21 - 45 years old.
* Within 4 months of a singleton, vaginal delivery

Exclusion Criteria:

* Currently pregnant
* Over 4 months since vaginal birth.
* Previous caesarean delivery.
* Previous pelvic floor surgery (eg. pelvic floor repair, continence surgery, cervicetomy,cosmetic pelvic floor procedures)
* Neurological disorder affecting muscle contraction (eg. Guillan-Barre syndrome, motorneuron disease, multiple sclerosis)

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Does visual feedback with transperineal ultrasound improve the effectiveness of pelvic floor muscle therapy in postpartum patients? | Baseline
  Is the change in antero-posterior pelvic hiatal diameter between rest and pelvic floor contraction better in the study arm compared to the control arm?

SECONDARY OUTCOMES:
Are postpartum patients who have trained with visual biofeedback more likely to continue to perform pelvic floor muscle therapy than those who do not train with visual biofeedback? | Baseline and 3 months later
  What is the reported change in frequency of pelvic floor contractions in the study group compared to the control group at the 3 month follow up?
Do postpartum patients who train with visual biofeedback continue to perform effective pelvic floor muscle contractions 3 months after pelvic floor muscle training | Baseline and at 3 months
  In the study group, is change in anteroposterior diameter maintained at the 3-month follow up?
Does pelvic floor contraction strength improve after 3 months of pelvic floor muscle therapy with visual biofeedback compared to those who did not receive visual biofeedback | Baseline and 3 months
  Does the change in antero-posterior pelvic hiatal diameter continue to be effective in the study group compared to the control group at the 3-month follow up?

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Obstetrics and Gynaecology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Consent to share IPD has not expressly been given by participants.

REFERENCES:
- [Background] Nyhus MO, Oversand SH, Salvesen O, Salvesen KA, Mathew S, Volloyhaug I. Ultrasound assessment of pelvic floor muscle contraction: reliability and development of an ultrasound-based contraction scale. Ultrasound Obstet Gynecol. 2020 Jan;55(1):125-131. doi: 10.1002/uog.20382. Epub 2019 Dec 13. PMID 31237722
- [Background] Frank DL, Khorshid L, Kiffer JF, Moravec CS, McKee MG. Biofeedback in medicine: who, when, why and how? Ment Health Fam Med. 2010 Jun;7(2):85-91. PMID 22477926
- [Background] Bo K, Owe KM, Nystad W. Which women do pelvic floor muscle exercises six months' postpartum? Am J Obstet Gynecol. 2007 Jul;197(1):49.e1-5. doi: 10.1016/j.ajog.2007.02.014. PMID 17618754
- [Background] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT07065708/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT07065708/ICF_001.pdf